CLINICAL TRIAL: NCT07024823
Title: A Phase I Randomized, Single-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD4248 Following Single and Multiple Ascending Dose Administration in Healthy Participants and Participants With Chronic Kidney Disease and Type 2 Diabetes and to Assess Home Measurements of Creatinine in a Prospective, Non-interventional Cohort Study
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD4248 in Healthy Participants and Participants With Chronic Kidney Disease and Type 2 Diabetes and to Assess Home Measurements of Creatinine in a Non Interventional Cohort
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D8380C00001
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease
Keywords: Type 2 Diabetes; Diabetic Kidney Disease; Multiple Ascending Dose; Single Ascending Dose; Creatinine; Food Effect; Pharmacokinetics; Safety
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A1 SAD (Experimental): Participants will receive single ascending oral dose of AZD4248 or placebo.
  Interventions: Drug: AZD4248; Drug: Placebo
- Part A2 SAD Chinese Cohort (Experimental): Participants will receive single oral dose of AZD4248 or placebo.
  Interventions: Drug: AZD4248; Drug: Placebo
- Part A3 SAD IV Cohort (Experimental): Participants will receive single IV infusion of AZD4248 or placebo.
  Interventions: Drug: AZD4248; Drug: Placebo
- Part B1 MAD (Experimental): Participants will receive multiple ascending oral doses of AZD4248 or placebo.
  Interventions: Drug: AZD4248; Drug: Placebo
- Part B2 MAD Japanese (Experimental): Participants will receive multiple ascending oral doses of AZD4248 or placebo.
  Interventions: Drug: AZD4248; Drug: Placebo
- Part C Multiple Dosing DKD (Experimental): Participants will receive multiple oral doses of AZD4248 or placebo.
  Interventions: Drug: AZD4248; Drug: Placebo
- Part D Observational Cohort (No Intervention): Participants will participate in home-based creatinine self-measurement.

INTERVENTIONS:
Drug: AZD4248 — AZD4248 will be administered orally.
  Arms: Part A1 SAD; Part A2 SAD Chinese Cohort; Part B1 MAD; Part B2 MAD Japanese; Part C Multiple Dosing DKD
Drug: Placebo — Placebo will be administered orally.
  Arms: Part A1 SAD; Part A2 SAD Chinese Cohort; Part B1 MAD; Part B2 MAD Japanese; Part C Multiple Dosing DKD
Drug: AZD4248 — AZD4248 will be administered via IV infusion.
  Arms: Part A3 SAD IV Cohort
Drug: Placebo — Placebo will be administered via IV infusion.
  Arms: Part A3 SAD IV Cohort

SUMMARY:
This study will evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending doses (SAD) and multiple ascending doses (MAD) of AZD4248 administered as an oral solution and intravenous (IV) infusion. Additionally, the study investigates the non-interventional feasibility of home measurement of serum creatinine in participants with diabetic kidney disease (DKD).

DETAILED DESCRIPTION:
This is a Phase I, first in human (FIH), randomized, single-blind, placebo-controlled study of AZD4248 involving healthy participants (Parts A and B) and participants with DKD (Part C) and to assess home measurements of creatinine in a prospective, non-interventional cohort in participants with DKD (Part D).

The study consists of 4 parts:

* Part A: SAD. Part A will consist of Parts A1 (single ascending doses in healthy participants), A2 (single dose in healthy Chinese participants), and A3 (IV infusion in healthy participants).
* Part B: MAD. Part B will consist of Parts B1 (multiple ascending doses in healthy participants) and B2 (multiple ascending doses in healthy participants of Japanese descent).
* Part C: Multiple dosing in participants with DKD.
* Part D: Multi-site, non-interventional, prospective cohort evaluation of home-based creatinine self-measurement in participants with DKD.

ELIGIBILITY:
Key Inclusion Criteria:

- Healthy participants with suitable veins for cannulation or repeated venipuncture.

Parts A and B:

* Have a body mass index (BMI) between 18 and 30 kilograms per millimeter (kg/m2), inclusive.
* For Chinese participants (Part A2): participants are to be Chinese, defined as having both parents and 4 grandparents who are Chinese. This includes second and third generation participants of Chinese descent whose parents or grandparents are living in a country other than China.
* For Japanese participants (Part B2): participants are to be Japanese, defined as having both parents and 4 grandparents who are Japanese. This includes second and third generation participants of Japanese descent whose parents or grandparents are living in a country other than Japan.

Part C:

* Have a BMI between 20 and 35 kg/m2, inclusive.
* Have a diagnosis of diabetic kidney disease (DKD).
* Hemoglobin A1C (HbA1c) of ≤ 10.5%.
* Participants are required to be on a stable dose of angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) for at least 6 weeks prior to Visit 1 and throughout the Screening Period. In addition, participants should be on stable doses of all other medication for ≥ 6 weeks before Screening.

Part D:

* Have a BMI between 20 and 35 kg/m2, inclusive.
* Have a diagnosis of DKD as defined by a) diagnosis of type 2 diabetes (T2D) b) eGFR values and c) urine albumin to creatinine ratio (UACR) values.
* HbA1c of ≤ 10.5%.
* Participants are required to be on a stable dose of ACEi or ARB for at least 6 weeks prior to Visit 1 and throughout the Screening Period. In addition, participants should be on stable doses of all other medication for ≥ 6 weeks before Screening.
* Participants must be able and motivated to use the home creatinine device and smartphone independently by successfully performing the test without assistance from site staff.
* Participants must be able to read and understand English sufficient to participate in site visits and home testing.

Key Exclusion Criteria:

* History of any clinically important disease or disorder which may put the participant at risk because of participation in the study or influence the results.
* Any positive result on Screening for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or human immunodeficiency virus (HIV).

Parts A and B:

* History or presence of gastrointestinal, hepatic, or renal disease.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4248.
* Participants who have previously received AZD4248.

Part C:

* History or presence of gastrointestinal, hepatic, or renal disease.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4248.
* Use of drugs that are strong or moderate CYP3A4 inhibitors/inducers or P-gp inhibitors from within 3 weeks before Screening until the end of the last sample collection.
* Participants who have previously received AZD4248.
* Participants on serum creatinine-altering drugs should be on long-term treatment at a stable dose prior to study entry.
* Expected change of dosing regimen during the study.
* History of clinically significant heart or vascular disease.
* New York Heart Association Class 2, 3, or 4 or history of hospitalization for heart failure within 6 months of screening.
* Ventricular arrhythmias requiring treatment.
* Amputation due to peripheral artery disease.
* Severe chronic obstructive pulmonary disease as judged by the Investigator or hospitalization for exacerbation in the last 6 months.

Part D:

* Participants on serum creatinine-altering drugs should be on long-term treatment at a stable dose prior to study entry.
* Expected change of dosing regimen during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Parts A, B, and C: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 to Follow Up visit (Part A: up to 12 days; Part B and C: up to 19 days)
  To assess the safety and tolerability of AZD4248 following single oral ascending doses or single IV administration to healthy participants and multiple oral ascending doses to healthy participants and participants with CKD and T2D (DKD).
Part D: Intra- and inter-participant variability of estimated glomerular filtration rate (eGFR) derived from home self-testing device measurements | Day 1 to Day 169
  To assess intra- and inter-participant variability of twice weekly home-based serum creatinine measurements.

SECONDARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
  To assess the impact of food on the PK of AZD4248 following a single oral administration.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
  To assess the impact of food on the PK of AZD4248 following a single oral administration.
Dose normalized AUClast (AUClast/D) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Dose normalized AUCinf (AUCinf/D) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Apparent total body clearance (CL/F) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Maximum observed drug concentration (Cmax) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
  To assess the impact of food on the PK of AZD4248 following a single oral administration
Dose normalized Cmax (Cmax/D) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Terminal elimination half-life (t½λz) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Terminal rate constant (λz) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Time delay between drug administration and the first observed concentration (tlag) | Part A1 and A2: Days 1-7, Part A3: Days 1-3.
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Time of last quantifiable concentration (tlast) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Time to reach maximum observed concentration (tmax) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
  To assess the impact of food on the PK of AZD4248 following a single oral administration
Apparent volume of distribution based on the terminal phase (Vz/F) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Absolute bioavailability (F) | Part A1 and A2: Days 1-7, Part A3: Days 1-3.
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Total body clearance (CL) | Part A1 and A2: Days 1-7, Part A3: Days 1-3, Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Volume of distribution at steady state (Vss) | Part A1 and A2: Days 1-7, Part A3: Days 1-3.
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Area under concentration-time curve in the dose interval (AUCtau) | Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Dose normalized AUCtau (AUCtau/D) | Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Accumulation ratio for AUC (Rac AUC) | Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV adnminstration of AZD4248.
Accumulation ratio for Cmax (Rac Cmax) | Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Temporal change parameter (TCP) | Part B: Days 1-17. Part C: Days 1-17
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248.
Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] | Part A: Days 1-2. Part B: Days 1-4 and 11-14. Part C: Days 1-4 and 11-14
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248
Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 [fe(t1-t2)] | Part A: Days 1-2. Part B: Days 1-4 and 11-14. Part C: Days 1-4 and 11-14
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248
Renal clearance (CLR) | Part A: Days 1-2. Part B: Days 1-4 and 11-14. Part C: Days 1-4 and 11-14
  To characterize the PK of AZD4248 following oral administration of single and multiple doses or a single IV administration of AZD4248
Percentage change from baseline in plasma target engagement marker | Part A: Days 1-5. Part B: Days 1-4 and 11-14. Part C: Days 1-4 and 11-14
  To evaluate the TE of AZD4248 by assessing reduction in plasma target engagement marker following single (oral or IV) and multiple oral dosing of AZD4248.
Part D: Intra- and inter-participant variability of eGFR derived from laboratory measurements | Day 1 to Day 169
  To assess the intra- and inter-participant variability of monthly laboratory-based creatinine measurements.
Part D: Changes over longitudinal follow-up in participant-reported experience questionnaire on collective participant satisfaction, usability and device acceptability data | Day 1 to Day 169
  To evaluate the usability, user satisfaction, and feasibility of delivering a home self-testing device and its accompanying smartphone application.
Part D: Summary of qualitative insights from optional individual in-depth interview samples | Day 30 to Day 84
  To evaluate the usability, user satisfaction, and feasibility of delivering a self-testing, home self-testing device and its accompanying smartphone application.
Part D: Changes over longitudinal follow-up in site-based staff reported PTSFQ | Day 1 to Day 169
  To assess clinical site staff-reported usability and satisfaction of delivering and management of the home self-testing device and software.
Part D: Estimated glomerular filtration rate (eGFR) | Day 1 to Day 169
  To compare home-based serum creatinine measurements against the standard laboratory measurements.
Part D: Proportion of completed creatinine tests, with completed assessments | Day 1 to Day 169
  To assess the rates of missing data due to missed tests or test errors.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Glendale, California
  - Research Site, Chicago, Illinois
  - Research Site, Ann Arbor, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/